CLINICAL TRIAL: NCT04134858
Title: The Effectiveness of Health Coaching for Frequent Attenders in the Primary Healthcare
Brief Title: The Effects of Health Coaching for Frequent Attenders
Acronym: HCFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Uoulu2014
Record Dates: First submitted 2019-09-16; First posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Health Behavior
Keywords: coaching; primary health care
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Intervention Model Description: The experimental and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The health coaching group (Experimental): The experimental group (n = 52) consisted of frequent attenders who had chosen the health-coaching program. The intervention was based on the customized nurse-led health-coaching program. The program consisted of an individual health-coaching nurse, health-coaching sessions and a written action plan according to each participant´s individual needs.
  Interventions: Other: The nurse-led health coaching program
- The control group (No Intervention): The control group consisted of 58 frequent attenders. They, along with the experimental group, received the usual care regarding their health problems from the physicians and nurses at the primary healthcare centres if they needed it. The usual care for frequent attenders included assessment for the need of treatment, physical examination, problem assessment, laboratory and X-ray tests, medical advice and patient support and education during their visits.

INTERVENTIONS:
Other: The nurse-led health coaching program — The intervention was based on the customized nurse-led health-coaching program. The program consisted of an individual health-coaching nurse, health-coaching sessions and a written action plan according to each participant´s individual needs.
  Arms: The health coaching group

SUMMARY:
The purpose of the study was to describe and evaluate the effectiveness of health coaching on health-related quality of life, adherence to health regimens, clinical health outcomes and lifestyle factors among frequent attenders in primary healthcare.

DETAILED DESCRIPTION:
The quasi-experimental research method evaluated the effectiveness of health coaching among frequent attenders in primary healthcare. The experimental group received the health coaching and the control group received the usual care. The data were collected with pre- and posttest 12-month follow-up via a questionnaire of FINRISKI2012, RAND-36 and ACDI and clinical health outcomes measured by health-coaching nurses. The data were analyzed by statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had face-to-face visits to the physicians in the local primary healthcare centre at least seven times during a 12-month period
* Aged 18 years or older
* Able to read and understand Finnish

Exclusion Criteria:

* Patients´ visits due to pregnancy or delivery
* Patients´ visits due to serial treatment for the same disease
* An inability to give informed consent
* Involving in another study intervention at the same time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2016-02-01 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
The health-related quality of life | 12 months
  The health-related quality of life was measured using the validated Finnish version of the RAND 36-Item Health Survey 1.0 (RAND-36). The 36-item self-report instrument consists of eight separate scales of quality of life: (1) physical functioning (10 items), (2) physical role functioning (four items), (3) emotional role functioning (three items), (4) social role functioning (two items), (5) bodily pain (two items), (6) mental health (five items), (7) energy (four items) and (8) general health (five items). The scores were calculated in a two-step process using the instructions provided by Ware et al. (1994) in the user´s manual. First, all items were scored on a scale from 0 to 100. A higher score defines a better health or function. Second, items in the same scale were averaged together to create the eight scale scores. Scale scores represented the average for all items in the scale.
Adherence to health regimens | 12 months
  Adherence was measured using the Adherence of People with Chronic Disease Instrument (ACDI) (Kyngäs, 1999), a 38-item self-report instrument that has been used to measure adherence to health regimens among people with chronic disease

SECONDARY OUTCOMES:
Lifestyle factors | 12 months
  The secondary outcomes were lifestyle factors. The baseline and follow-up questionnaires gathered data on the frequent attenders' alcohol consumption, smoking behaviour, and physical activity. They were based on a customized variant of the national FINRISK 2012 questionnaire

OTHER OUTCOMES:
The clinical health outcomes: Weight | 12 months
  Weight in kilograms (kg)
The clinical health outcomes: Height | 12 months
  Height in meters (m)
The clinical health outcomes: Body mass index (BMI) | 12 months
  Weight and height will be combined to report BMI in kg/m^2
The clinical health outcomes: Blood pressure | 12 months
  Blood pressure were measured using systolic and diastolic blood pressure in mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Kääriäinen, Professor, Study Director — University of Oulu

IPD SHARING:
Plan to Share IPD: No